CLINICAL TRIAL: NCT05105191
Title: Analytical Performances and Clinical Impact of the Roche Cobas® Liat Influenza A/B & RSV Assay in the Management of Adult and Pediatric Patients Attending the Emergency Room
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic introduced a confusion bias
Sponsor: Erasme University Hospital (Other)
Collaborators: LHUB-ULB (Unknown); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SRB2019_401
Record Dates: First submitted 2021-09-29; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Influenza Viral Infections; RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Roche Cobas® Liat Influenza A/B & RSV assay — Performance of a rapid molecular assay to diagnose influenza and RSV infections

SUMMARY:
Molecular techniques for respiratory virus detection have already shown benefits in terms of sensitivity gained in comparison to conventional techniques. Recent progress has made it possible to shorten turnaround time (TAT) and to allow delivery of results in a timely manner, especially in comparison to cell culture and direct fluorescence assays (DFA). However, the cost of these molecular assays is usually not taken in charge by public health insurance system. This could be partly explained by the fact that molecular techniques have not clearly shown cost-effectiveness. Results of molecular tests for influenza viruses and RSV, if delivered rapidly, in the emergency room (ER), would most likely help avoid antibiotic use and ancillary test prescription, improve antiviral prescription and shorten length of stay in the ward by facilitating discharge or cohorting of hospitalized patients. The goal of this study is to assess the performances of Roche Cobas® Liat Influenza A/B & RSV assay, to appraise its clinical impact and to evaluate its cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Either a pre-test indication of hospitalization
* or an underlying situation at risk of respiratory complication following influenza infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Analytical performance (Sensitivity/Specificity) | through study completion, 6 months
  Calculation of sensitivity and specificity of the test versus a composite reference standard. Samples are considered as positive for a viral pathogen if testing positive for this viral pathogen by at least 2 of the 3 techniques used, negative if tested negative by at least 2 of the 3 techniques (culture, antigen detection and PCR test).
Hospital admission intentions | through study completion, 6 months
  Number of admission intentions before and after the test result
Isolation intentions | through study completion, 6 months
  Number of isolation intentions before and after the test result
Antibiotic prescription intentions | through study completion, 6 months
  Number of antibiotic prescription intentions before and after the test result
Antiviral treatment prescription intentions | through study completion, 6 months
  Number of antiviral treatments prescription intentions before and after the test result

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - Brugmann Hospital, Brussels
  - Erasme Hospital, Brussels
  - HUDERF, Brussels
  - Saint-Pierre Hospital, Brussels